CLINICAL TRIAL: NCT05753631
Title: Evaluation of the Effects of Injectable Platelet-rich Fibrin (i-PRF) Application on Periodontal Clinical and Biochemical Parameters in Gingival Crevicular Fluid (GCF) in Non-surgical Periodontal Treatment
Brief Title: Effects of i-PRF on Non-surgical Periodontal Treatment
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, AYSAN LEKTEMUR ALPAN, Associate Profesor, Pamukkale University
Other Study IDs: 22.02.2022/04
Record Dates: First submitted 2023-01-18; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Platelet-Rich Fibrin
Keywords: platelet-rich fibrin; non-surgical periodontal treatment; wound healing; growth factor; cytokine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SRP+i-PRF (test): Injectable platelet-rich fibrin (i-PRF) application into the selected deep periodontal pocket after scaling and root planning (SRP) procedure.
  Interventions: Procedure: non surgical periodontal treatment
- SRP (Control): No agent was applied to the periodontal pocket after scaling and root planning.
  Interventions: Procedure: non surgical periodontal treatment

INTERVENTIONS:
Procedure: non surgical periodontal treatment — scaling and root planning were applied for non-surgical periodontal treatment i-PRF application: Intravenous blood sample taken from the antecubital vein of the patients was collected in a 10 ml tube and centrifuged at 700 rpm for 3 minutes in a PRF centrifuge device. The PRF obtained from the upper liquid layer formed in the tube was injected subgingival into the deepest point of the pocket after SRP treatment.
  Clinical periodontal measurements: plaque index, gingival index, probing depth, clinical attachment level, bleeding on probing, and gingival recession were calculated.
  gingival crevicular fluid: Perio papers were placed in the deepest part of the sulcus and left for 30 seconds. After 30 seconds, the paper strips were placed in the periotron device and the volume was calculated.
  Other Names: i-PRF application; clinical periodontal measurement taken; gingival crevicular fluid obtained

SUMMARY:
Injectable platelet-rich fibrin, a platelet concentrate in a liquid formulation, has been developed to provide clinicians with ease of use alone or in combination with various biomaterials. The low-speed centrifugation method provides a significant advantage to the regeneration process with richer platelets, leukocytes, and growth factors. It also contributes to the wound-healing process by increasing vascularization. It is expected that the application of injectable platelet-rich fibrin into the gingival pocket following subgingival curettage in periodontitis patients will positively affect the results of non-surgical periodontal treatment. For this reason, in this study it was aimed to investigate the early effects of injectable PRF applied into the pocket for root surface biomodification following subgingival curettage in periodontal pockets of 6 mm and above, by evaluating both clinical parameters and inflammatory and healing markers in the gingival groove fluid

DETAILED DESCRIPTION:
The study was planned as a randomized controlled split-mouth clinical trial. A split-mouth design was used to better assess how the same host responded to two different treatment modalities. Two quadrants with contralateral deep periodontal pockets in each participant were selected and randomly divided into test and control groups.

Test group: Injectable platelet-rich fibrin application into the selected deep periodontal pocket after scaling and root planning (SRP) procedure.

Control group: No agent was applied to the periodontal pocket after scaling and root planning.

On the first visit, clinical periodontal measurements were taken before the SRP procedure. Plague index (PI), gingival index (GI), probing depth (PD), clinical attachment level (CAL), and bleeding on probing (BOP) were used as clinical periodontal parameters.

After 1 week, the patients were called again for the SRP procedure. Injectable PRF obtained from the intravenous blood sample taken from the antecubital vein of the patients was injected into the deepened periodontal pocket subgingivally after the SRP procedure in the test group. Clinical periodontal measurements at 1 month and 3 months after SRP were repeated.

Gingival crevicular fluid (GCF) samples were taken from selected teeth before the SRP procedure. On the 3rd and 7th day after the SRP, GCF samples were taken again from the same region.

GCF vascular endothelial growth factor (VEGF), tumor necrosis factor-alpha (TNF-α), and interleukin (IL)-10 levels were evaluated by using the ELISA method and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* patients with stage 3 grade B periodontitis

Exclusion Criteria:

* patients with systemic disease
* pregnant and breastfeeding
* acute or chronic infection in the past 6 months
* Use of systemic antibiotic therapy in the past 6 months
* use of drugs that can affect periodontal health
* receiving hormone therapy
* smokers
* teeth with endodontic lesions
* Teeth with class 2 and 3 mobility

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemically healthy and stage 3 grade B periodontitis aged 18-65
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
GCF VEGF levels in test and control groups | Change from Baseline GCF VEGF levels at 3rd and 7th days
  measure and compare the improvement of VEGF in test and control groups by using ELISA
GCF TNF-alpha levels in test and control groups | Change from Baseline GCF TNF-alpha levels at 3rd and 7th days
  measure and compare the improvement of TNF-alpha in test and control groups by using ELISA
GCF IL-10 levels in test and control groups | Change from Baseline GCF IL-10 levels at 3rd and 7th days
  measure and compare the improvement of IL-10 in test and control groups by using ELISA
Plaque index (PI) | Change from Baseline PI at 3rd and 7th days
  measure and compare the improvement of PI in test and control groups using a scale
Probing depth (PD) | Change from Baseline PD levels at 3rd and 7th days
  measure the gingival margin to pocket bottom as mm and compare the improvement of PD in test and control groups
Gingival index (GI) | Change from Baseline GI at 3rd and 7th days
  measure and compare the improvement of GI in test and control groups using a scale
Bleeding on probing (BOP) | Change from Baseline BOP at 3rd and 7th days
  Whether there is bleeding when the periodontal pocket is probed and comparing the improvement in test and control groups
Clinical attachment level (CAL) | Change from Baseline CAL at 3rd and 7th days
  measure the distance from the cemento-enamel line to the bottom of the pocket and compare the improvement in test and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Torumtay Cin, PhD, Principal Investigator — pamukkale university faculty of dentistry
Locations (1):
- Gizem Torumtay Cin, Denizli, Deni̇zli̇, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is planned to be given if requested with a valid reason.

REFERENCES:
- [Background] Miron RJ, Fujioka-Kobayashi M, Hernandez M, Kandalam U, Zhang Y, Ghanaati S, Choukroun J. Injectable platelet rich fibrin (i-PRF): opportunities in regenerative dentistry? Clin Oral Investig. 2017 Nov;21(8):2619-2627. doi: 10.1007/s00784-017-2063-9. Epub 2017 Feb 2. PMID 28154995
- [Result] Choukroun J, Diss A, Simonpieri A, Girard MO, Schoeffler C, Dohan SL, Dohan AJ, Mouhyi J, Dohan DM. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part IV: clinical effects on tissue healing. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e56-60. doi: 10.1016/j.tripleo.2005.07.011. PMID 16504852
- [Derived] Torumtay Cin G, Lektemur Alpan A, Cevik O. Efficacy of injectable platelet-rich fibrin on clinical and biochemical parameters in non-surgical periodontal treatment: a split-mouth randomized controlled trial. Clin Oral Investig. 2023 Dec 28;28(1):46. doi: 10.1007/s00784-023-05447-8. PMID 38153510